CLINICAL TRIAL: NCT05083637
Title: Role of L-Carnitine Supplementation on Rate of Weight Gain and Biomarkers of Environmental Enteric Dysfunction (EED) in Children With Severe Acute Malnutrition
Brief Title: L-Carnitine Supplementation, Rate of Weight Gain and EED in Children With SAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PR-21046
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-01

CONDITIONS: Malnutrition
Keywords: Malnutrition; L-Carnitine; Environmental Enteric Dysfunction; Under-5 children; Bangladesh
MeSH Terms: conditions — Malnutrition | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Active Comparator): Children randomized to this arm will receive L- carnitine oral solution (100mg/ml) (Generic Name) with the dosage- 100 mg/kg/day, divided into 3 doses per day for 15 days.
  Interventions: Drug: L- carnitine oral solution
- Control Arm (Placebo Comparator): Children randomized to this arm will receive placebo in same quantity, divided into 3 doses per day for 15 days.Placebo solution will be identical in appearance, smell and taste to the active preparation (L-carnitine syrup) with no therapeutic value.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L- carnitine oral solution — The L-carnitine syrup formulation will be provided to study participant at nutritional rehabilitation unit (NRU) under controlled set-up
  Other Names: Levocarnitine oral solution
  Arms: Intervention Arm
Other: Placebo — The placebo formulation will be provided to study participant at nutritional rehabilitation unit (NRU) under controlled set-up
  Arms: Control Arm

SUMMARY:
Background:

Burden:

Globally, an estimated 14.3 million under-5 children are severely malnourished. Two-thirds of them live in Asian countries, including Bangladesh. Acute malnutrition is an underlying cause of nearly half of global deaths in under-5 children despite standardized rehabilitation protocols. It is also associated with high relapse rates following discharge.

Knowledge Gap:

Malnourished children suffer from deficiencies of several essential nutrients. Studies showed that malnourished children had lower serum carnitine levels and demonstrated its role in the rate of weight gain in children with severe acute malnutrition (SAM). The consequences of nutritional impairment can be perilous if carnitine deficiency is coupled with Environmental Enteric Dysfunction (EED). Recent evidence confirms that EED is characterized by secondary carnitine deficiency in children. Carnitine deficiency leading to EED may cause childhood growth faltering and impaired cognitive development. However, evidence on carnitine status and its consequences in relation to EED in diarrheal children with SAM is very limited in Bangladesh.

Relevance:

Such lack of information regarding the role of L-carnitine in improving the rate of weight gain in malnourished children susceptible to EED is an obstacle in limiting the relapse and adverse consequences of SAM in diarrheal children living in resource-limited countries.

Hypothesis: L- carnitine supplementation for 15 days in children with SAM will improve the rate of weight gain and biomarkers of EED

Objective:

1. To investigate the role of L-carnitine supplementation on the rate of weight gain among the children with SAM
2. To investigate the role of L-carnitine supplementation on the duration of the hospital stays
3. To examine the role of L-carnitine supplementation on EED biomarkers, for instance, myeloperoxidase (MPO), neopterin (NEO), alpha-1 anti-trypsin (A1AT), kynurenine: tryptophan (KT) ratio, and citrulline in children with SAM

Methods: This study will be a double-blinded, placebo-controlled randomized clinical trial

DETAILED DESCRIPTION:
Study Design:

Study Site:

This study will be done in the Dhaka Hospital at icddr,b.

Study population:

In this study, the investigator will enroll diarrheal children with SAM aged 9-24 months of both genders attending longer stay units (LSU).

Study duration: 12 months

Screening, Consenting, and Baseline Data Collection:

The research staff ( Field Research Assistant) will screen all the participants within the defined age groups according to the eligibility criteria (Detailed inclusion/exclusion criteria are provided separately below). Then research staff will explain the study in detail, answer any questions from the parent(s), and invite the parent(s) to enroll the child in the study. If the parent(s) are interested in volunteering in the study, the designated staff will proceed to consent consisting of a thorough review of the written consent form in a manner appropriate for the child's parents' literacy level. Prior to signing the consent form, parent(s) will have an opportunity to ask any questions about the study participants fulfilling the eligibility criteria will be brought to the study physician for clinical assessment. If the parent(s) are not sufficiently literate to read and/or sign the consent form, consenting and fingerprint signature will be obtained in the presence of a witness who is not associated with the study. The child's parent(s) will be provided with a copy of the signed consent form. Upon signing a written informed consent, the participant will be enrolled by the study physician.

Randomization:

Participants will be assigned to the intervention or the control arm using permuted block randomization method with concealment to ensure that the allocation is not made before the participant has given their consent and joined the study. A random allocation sequence will be generated using a computerized random allocation system for permuted block randomization to ensure comparable allocation numbers at certain equally spaced points in the sequence of patient assignments. A parallel type of randomization will be used. Reasonably large blocks with variable block sizes will be constructed to reduce the predictability. Random assignment will be prepared in advance by an independent researcher from icddr,b, who has no involvement with the trial.

Anthropometric measurements:

All the measurements will be taken at enrollment and each day when the participants will receive intervention/placebo. End-line anthropometry data will be collected on the 15th day of supplementation. In addition, we will measure anthropometry on the 180th day after the completion of supplementation to observe the long-term effect of the intervention on the rate of weight gain. Trained staff will take all the measures as per the standard operating procedures (SOPs) and keep records in standard CRFs. The Seca weighing scale will be used for weight measurement in kg, and the Seca length board will be used for length measurement in cm. And mid-upper arm circumference (MUAC) will be measured in cm using a non-stretch tape.

Intervention:

The intervention will be given to the child along with the standard of treatment at the nutritional rehabilitation unit (NRU). Detailed information about the investigational product is provided separately below. Children will be monitored daily by trained physicians for any side effects/adverse events (such as nausea, vomiting, diarrhea, rash, urticaria, or any significant changes in clinical status). If any adverse events are observed, children will be treated using appropriate management practices at Dhaka Hospital.

Biological sample collection:

The investigators will collect blood, stool, and urine from the participants at enrolment and at the end of the nutrition intervention. Overall, 5 ml of whole venous blood will be collected aseptically from each of the participants as per the SOPs. The blood biomarkers that will be tested in this study are L-carnitine, Citrulline, KT Ratio, C-reactive protein (CRP), and Alpha-1-acid glycoprotein (AGP). CRP is an acute-phase protein and can be detected during infection. Increased level of AGP in serum indicates systemic tissue injury, inflammation, and infection. Both Citrulline and KT ratios indicate EED in children. The stool will be collected to investigate the concentrations of MPO, NEO, and A1AT in the fecal samples. The investigators will measure L-carnitine levels in the urine samples of each participant. All the assays will be done at icddr,b.

Laboratory Investigation:

The investigators will measure L-carnitine levels in plasma and urine and EED biomarkers in every enrolled patient. Pre and post-test will be done. The pre-test will be on the first day of enrolment, and the post-test will be on the 15th day after the completion of supplementation.

Sample Size Calculation:

The sample size is estimated considering the primary outcome variable. For the primary objective, the investigators have considered an intervention study in Turkey. The study discovered that the mean difference between the rate of weight gain in malnourished children after L-carnitine supplementation was 2.4 (The weight was measured in kg) with a standard deviation of 4.3. Setting the level of confidence at 95% (Z1-α =1.645) and the study power at 80%, the estimated sample size is 49 participants in each group with a 10% attrition rate. So, the total sample size for this study will be 98.

Data Analysis Plan:

Data will be entered into the pre-tested case record forms (CRFs) using Statistical Package for the Social Sciences (SPSS 20.0 version) and finally cleaned with a repeated check. Data will be presented using frequency with percentages for categorical variables. Mean with standard deviation will be used for symmetrical continuous variables. Median with interquartile range will be used for asymmetrical numeric variables. To know the outcome of the intervention in our study children bivariate, crude analyses of the association will be done that will involve Chi-square or Fisher's exact test for comparing differences in proportion and t-tests for numeric variables between the groups. Nonparametric continuous data will be analyzed by Mann-Whitney U-test. Results from all children will be included in the analysis of the study on an intention-to-treat basis. Data from children withdrawn because of failure to respond, or voluntary dropouts will be included in the analysis up to the time of withdrawal. A supplementary analysis excluding the children withdrawn may also be done. A probability of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diarrheal children with SAM aged 9-24 months
* Signed informed consent by the guardian/caregivers

Exclusion Criteria:

* Severe sepsis or Septic shock
* Patients already taking medications containing L- carnitine
* Children with Tuberculosis
* Children with congenital defects or chromosomal anomalies
* Children with a diagnosed case of Thalassemia
* Children with an active or previous history of convulsion

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of weight gain | Baseline to 15th day of treatment
  The rate of weight gain (g/kg/day) will be calculated by using the formulae below:
  [{Weight on completion of study - Weight on enrolment (or at no edema) (g)} / {Total duration (in days) * weight on enrolment in kg}]

SECONDARY OUTCOMES:
Duration of hospital stays | Baseline to 15 days of treatment
  It will be assessed by comparing duration of total hospital stay between the two arm
EED biomarkers [myeloperoxidase (MPO), neopterin (NEO), alpha-1 anti-trypsin (A1AT), kynurenine: tryptophan (KT) ratio, and citrulline] | Baseline to 15 days of treatment
  Biological sample will be analyzed using ELISA- based measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jinat Alam, MBBS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital; International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
After the end of the study, data will be analyzed as per the defined data analysis plan on the protocol. Study results will be shared with other researchers by journal publications, conferences proceedings, and dissemination programs

REFERENCES:
- [Background] Alp H, Orbak Z, Akcay F, Tan H, Aksoy H. Plasma and urine carnitine levels and carnitine supplementation in children with malnutrition. J Trop Pediatr. 1999 Oct;45(5):294-6. doi: 10.1093/tropej/45.5.294. PMID 10584472
- [Derived] Alam J, Fahim SM, Islam MR, Alam MA, Gazi MA, Ahmed T. Effects of L-Carnitine Supplementation on the Rate of Weight Gain and Biomarkers of Environmental Enteric Dysfunction in Children with Severe Acute Malnutrition: A Double-Blind Randomized Controlled Clinical Trial. J Nutr. 2024 Mar;154(3):949-961. doi: 10.1016/j.tjnut.2024.01.031. Epub 2024 Feb 6. PMID 38331348
- [Derived] Alam J, Islam MR, Fahim SM, Gazi MA, Ahmed T. Role of L-Carnitine supplementation on rate of weight gain and biomarkers of Environmental Enteric Dysfunction in children with severe acute malnutrition: A protocol for a double-blinded randomized controlled trial. PLoS One. 2022 Sep 30;17(9):e0275291. doi: 10.1371/journal.pone.0275291. eCollection 2022. PMID 36178918